CLINICAL TRIAL: NCT05774028
Title: A Single-arm, Multi-center Phase II Clinical Study on Pegaspargase Combined With Gemcitabine, Etoposide, Liposomal Mitoxantrone Hydrochloride and Dexamethasone (P-GEMD) in the Treatment of Untreated Early Non-upper Respiratory Tract or Advanced Extranodal NK/T-cell Lymphoma.
Brief Title: Pegaspargase Combined With Gemcitabine, Etoposide, Liposomal Mitoxantrone Hydrochloride and Dexamethasone (P-GEMD) in the Treatment of Untreated Early Non-upper Respiratory Tract or Advanced Extranodal NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-SR-002
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: NK-T-Cell Lymphoma, Extranodal
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Gemcitabine; Etoposide; Dexamethasone; Clinical Protocols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P-GEMD group (Experimental): Pegaspargase Combined With Gemcitabine, Etoposide, Liposomal Mitoxantrone Hydrochloride and Dexamethasone (P-GEMD) regimen
  Interventions: Drug: Pegaspargase Combined With Gemcitabine, Etoposide, Liposomal Mitoxantrone Hydrochloride and Dexamethasone (P-GEMD) regimen

INTERVENTIONS:
Drug: Pegaspargase Combined With Gemcitabine, Etoposide, Liposomal Mitoxantrone Hydrochloride and Dexamethasone (P-GEMD) regimen — P-GEMD regimen (Every 3 weeks as a cycle, a total of 6 cycles) : Pegaspargase 3750 IU, d2; Gemcitabine 1000mg/m2, d1; Etoposide 65mg/m2, d2-d4; Mitoxantrone hydrochloride liposome 12mg/m2, d1; Dexamethasone 40mg/d, d1- d4.

SUMMARY:
NK/T-cell lymphoma (NKTCL) is one of the most common types of extranodal lymphoma.NKTCL originates from NK cells and T lymphocytes and is highly invasive. There is a lack of efficient and specific treatment methods in clinical practice, and the prognosis is poor. The molecular heterogeneity of NKTCL is strong, and molecular typing and risk stratification are of great significance for understanding the disease and improving the curative effect.Based on the preclinical studies of mitoxantrone liposomes, the investigators put forward a hypothesis: mitoxantrone liposome injection combined with pegaspargase, gemcitabine, and dexamethasone (P-GEMD) in the treatment of early non-upper respiratory digestive tract It is safe and can improve the therapeutic effect in patients with gastric or advanced extranodal NK/T cell lymphoma.

DETAILED DESCRIPTION:
NK/T-cell lymphoma (NKTCL) is one of the most common types of extranodal lymphoma.NKTCL originates from NK cells and T lymphocytes and is highly invasive. There is a lack of efficient and specific treatment methods in clinical practice, and the prognosis is poor. The molecular heterogeneity of NKTCL is strong, and molecular typing and risk stratification are of great significance for understanding the disease and improving the curative effect.

In the phase II clinical study of mitoxantrone liposome, 108 patients with relapsed and refractory PTCL received mitoxantrone liposome monotherapy, and the IRC evaluation ORR was 41.7% [32.3%, 51.5%] , the CR rate was 23.1% (25/108), the median PFS was 8.5 months, and the median OS was 22.8 months. The safety was tolerable and the efficacy was definite. Based on this, Mitoxantrone liposome was approved for marketing , for the treatment of adult patients with relapsed and refractory PTCL.

Based on the preclinical studies of mitoxantrone liposomes, the investigators put forward a hypothesis: mitoxantrone liposome injection combined with pegaspargase, gemcitabine, and dexamethasone (P-GEMD) in the treatment of early non-upper respiratory digestive tract It is safe and can improve the therapeutic effect in patients with gastric or advanced extranodal NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily join this study and sign the informed consent form; 2. 18 years old ≤ age ≤ 75 years old; 3. Expected survival time ≥ 3 months; 4. Histopathologically confirmed early non-upper aerodigestive or advanced 5. There must be at least one evaluable or measurable lesion that meets the Lugano2014 criteria: lymph node lesions, measurable lymph nodes need to have a long diameter > 1.5cm; non-lymph node lesions, extranodal lesions that can be measured Long diameter > 1.0cm; 6. ECOG score 0-2 points; 7. Bone marrow function: neutrophil count ≥ 1.5×109/L, platelet count ≥ 75×109/L, hemoglobin ≥ 80g/L; 8. Liver and kidney function: serum creatinine ≤ 1.5 times the upper limit of the normal value; alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5 times the upper limit of the normal value (for patients with liver invasion ≤ 5 times the normal value upper limit); total bilirubin ≤ 1.5 times the upper limit of normal value (for patients with liver invasion ≤ 3 times the upper limit of normal value).

Exclusion Criteria:

* 1. Hypersensitivity to any study drug or its components; 2. Uncontrollable systemic diseases (such as advanced infection, uncontrollable hypertension, diabetes, etc.); 3. Cardiac function and disease meet one of the following conditions :

  1. long QTc syndrome or QTc interval >480 ms;
  2. complete left bundle branch block, second-degree or third-degree atrioventricular block;
  3. severe, uncontrolled arrhythmia requiring drug treatment ;
  4. New York Society of Cardiology ≥ Grade III;
  5. Cardiac ejection fraction (LVEF) lower than 50%;
  6. Myocardial infarction, unstable angina, and severely unstable ventricular rhythm within 6 months before recruitment History of arrhythmia or any other arrhythmia requiring treatment, history of clinically severe pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities.

     4. Active hepatitis B and C infection (positive hepatitis B virus surface antigen and more than 1x103 copies/mL of hepatitis B virus DNA; more than 1x103 copies/mL of hepatitis C virus RNA); 5. Human immunodeficiency virus (HIV) infection (positive HIV antibody); 6. Previously or currently suffering from other malignant tumors (except for effectively controlled non-melanoma skin basal cell carcinoma, breast/cervix carcinoma in situ and other malignant tumors that have been effectively controlled without treatment in the past five years); 7. Central nervous system (CNS) involvement at the time of recruitment; 8. Pregnant, lactating women and patients of childbearing age who do not want to take contraceptive measures; Other investigators judge that they are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
CRR | 6 months
  Complete Response Rate

SECONDARY OUTCOMES:
ORR | 6 months
  Objective Response Rate
DoR | 1 years
  Duration of remission
1 year PFS rate | 1 years
  1 year PFS rate
1 year OS rate | 1 years
  1 year OS rate